CLINICAL TRIAL: NCT01434953
Title: Diagnostic Labeling: Effect on White Coat Hypertension
Brief Title: Prehypertension Labeling
Acronym: Tanya K23
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAAC6382
Record Dates: First submitted 2011-09-08; First posted 2011-09-15 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Prehypertension
Keywords: Prehypertension; Blood pressure screening; White coat effect
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Labeled (Experimental)
  Interventions: Behavioral: Labeled prehypertension
- Unlabeled (Active Comparator)
  Interventions: Behavioral: Unlabeled prehypertension

INTERVENTIONS:
Behavioral: Labeled prehypertension — A study physician informs subjects of their blood pressure level. Subjects are told they have prehypertension and are informed of the associated health risks.
  Arms: Labeled
Behavioral: Unlabeled prehypertension — A study physician informs subjects of their blood pressure level. The term "prehypertension" is not used and associated health risks are not discussed.
  Arms: Unlabeled

SUMMARY:
The purpose of this study is to find out whether labeling adults with prehypertension has negative effects on clinic blood pressure and quality of life 3 months after diagnosis.

DETAILED DESCRIPTION:
Previous research has shown that a diagnosis of hypertension is associated with subsequent increases in resting blood pressure, and there is preliminary evidence of a cross-sectional association between hypertension labeling and the white coat effect. The white coat effect may be particularly problematic in prehypertensives, because a small elevation in clinic blood pressure could result in crossing the diagnostic cutoff for hypertension, potentially leading to misdiagnosis and unnecessary treatment. This study will examine effects of prehypertension labeling on clinic and ambulatory blood pressure, and will examine potential psychological mediators of these associations.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* average screening systolic blood pressure of 120-139 mmHg OR diastolic blood pressure of 80-89 mmHg
* average screening systolic blood pressure below 140 mmHg AND diastolic blood pressure below 90 mmHg
* able to read and write in English

Exclusion Criteria:

* past diagnosis of hypertension, prehypertension, or high blood pressure
* current or past use of antihypertensive medications
* diabetes
* renal disease
* cardiovascular disease
* current participation in another hypertension-related clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07-13 (Actual); Primary Completion 2012-07-09 (Actual); Study Completion 2012-07-09 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline, 3 months

SECONDARY OUTCOMES:
Change in health-related quality of life (SF-12 questionnaires) | Baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Burg, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States